CLINICAL TRIAL: NCT04943848
Title: A Phase I Clinical Trial of Neo-antigen Heat Shock Protein Vaccine (rHSC-DIPGVax) in Combination With Checkpoint Blockade for the Treatment of Diffuse Intrinsic Pontine Glioma (DIPG) and Diffuse Midline Glioma in Childhood
Brief Title: rHSC-DIPGVax Plus Checkpoint Blockade for the Treatment of Newly Diagnosed DIPG and DMG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Children's Hospital of Orange County (Other); University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LCH 20C05
Record Dates: First submitted 2021-05-24; First posted 2021-06-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant
Keywords: Immunotherapy; Cancer vaccine; Checkpoint blockade; DIPG; Diffuse intrinsic pontine glioma; High grade glioma; DMG; Diffuse midline glioma; rHSC-DIPGVax; Balstilimab; Zalifrelimab
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Vaccines; balstilimab; Immune Checkpoint Inhibitors; spartalizumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Phase I, open label, plus expansion clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- "Lead In": rHSC-DIPGVax Monotherapy (Experimental): rHSC-DIPGVax for 8 total doses
  Interventions: Biological: rHSC-DIPGVax
- Part A: rHSC-DIPGVax in Combination with BALSTILIMAB (Anti-PD1) (Experimental): rHSC-DIPGVax (8 total doses) + BALSTILIMAB (1 year of therapy or 27 cycles, whichever comes first)
  Patients will enroll 6-10 weeks post standard of care (SOC) radiation completion. Steroid dose must be at or below 0.5mg/kg/day for a minimum of 7 days. The first 3 patients must be 5 years or older to 18. Subsequently, subjects ages 12 months to 18 years can be enrolled. Up to six patients will be enrolled on Part A. Once safety is established for rHSC-DIPGVax plus anti-PD1 (BALSTILIMAB), the study will proceed to Part B.
  Interventions: Biological: rHSC-DIPGVax; Drug: Balstilimab
- Part B: Dose Escalation of ZALIFRELIMAB (Anti-CTLA4) (Experimental): rHSC-DIPGVax (8 total doses) + BALSTILIMAB + ZALIFRELIMAB (1 year of therapy or 9 cycles, whichever comes first)
  Patients will enroll 6-10 weeks post standard of care (SOC) radiation therapy. Steroid dose must be at or below 0.5mg/kg/day for a minimum of 7 days. The first 3 patients must be 5 years or older to 18. Subsequently, subjects ages 12 months to 18 years can be enrolled. Up to 12 patients will be enrolled on Part B. Once safety is established for rHSC-DIPGVax plus anti-PD1 (BALSTILIMAB) plus anti-CTLA4 (ZALIFRELIMAB), the study will proceed to Part C.
  Interventions: Biological: rHSC-DIPGVax; Drug: Balstilimab; Drug: Zalifrelimab
- Part C: Dose Expansion (Experimental): rHSC-DIPGVax (8 total doses) + BALSTILIMAB + ZALIFRELIMAB (at RP2D from Part B) (1 year of therapy or 9 cycles, whichever comes first)
  Patients will enroll 6-10 weeks post standard of care (SOC) radiation therapy. Steroid dose must be at or below 0.5mg/kg/day for a minimum of 7 days. Up to 12 patients will be enrolled on Part C. All subjects in Part C will be monitored for DLT's for the duration of their participation in the study to monitor for excess toxicity.
  Interventions: Biological: rHSC-DIPGVax; Drug: Balstilimab; Drug: Zalifrelimab

INTERVENTIONS:
Biological: rHSC-DIPGVax — Off-the-shelf, neoantigen heat shock protein vaccine
  Other Names: vaccine
Drug: Balstilimab — BALSTILIMAB is a human monoclonal antibody that targets programmed cell death 1 (PD1)
  Other Names: checkpoint blockade; anti-PD1
  Arms: Part A: rHSC-DIPGVax in Combination with BALSTILIMAB (Anti-PD1); Part B: Dose Escalation of ZALIFRELIMAB (Anti-CTLA4); Part C: Dose Expansion
Drug: Zalifrelimab — ZALIFRELIMAB is a human monoclonal immunoglobulin G1k subclass (IgG1k) antibody that specifically recognizes cytotoxic T lymphocyte-associated protein 4 (CTLA-4, also known as CD152)
  Other Names: checkpoint blockade; anti-CTLA4
  Arms: Part B: Dose Escalation of ZALIFRELIMAB (Anti-CTLA4); Part C: Dose Expansion

SUMMARY:
This is a phase I, open label, plus expansion clinical trial evaluating the safety and tolerability of rHSC-DIPGVax in combination with BALSTILIMAB and ZALIFRELIMAB. rHSC-DIPGVax is an off-the-shelf neo-antigen heat shock protein containing 16 peptides reflecting neo-epitopes found in the majority of DIPG and DMG tumors. Newly diagnosed patients with DIPG and DMG who have completed radiation six to ten weeks prior to enrollment are eligible.

DETAILED DESCRIPTION:
This is a phase I, open label, plus expansion clinical trial evaluating the safety and tolerability of rHSC-DIPGVax in combination with BALSTILIMAB and ZALIFRELIMAB using a 3+3 design for subjects with newly diagnosed DIPG or DMG following completion of radiation therapy. Given this is a first in-human study of rHSC-DIPGVax, an initial study "Lead In" will assess the tolerability of vaccine monotherapy first in older children (ages 5 to 18 years of age) followed by younger children (12 months to 18 years of age).

Sequential Parts A and B of this study will also first enroll patients ages 5 to 18 years of age before enrolling younger children. The rationale for the combination of vaccine and anti-PD1 therapy includes evidence of a more profound intra-tumoral response with addition of inhibition of negative co-regulatory pathways, such as, PD1/PDL1 and the need to overcome potentially immunosuppressive or immune "cold" microenvironment of gliomas. Anti-CLTA4 therapy will also be combined with rHSC-DIPGVax in the dose escalation portion of this study because of the ability of anti-CTLA4 therapy to induce T cell priming to promote T memory formation. Given the lack of standard treatment options for DIPG and DMG patients, this clinical trial will use combinatorial immunotherapy in upfront treatment of these patients in hopes of maximizing potential efficacy in this at-risk population while still assessing safety throughout.

Part A will evaluate rHSC-DIPGVax plus BALSTILIMAB. Pharmacokinetics (PK) of BALSTILIMAB will also be evaluated to assess exposure. If the rHSC-DIPGVax plus BALSTILIMAB is well tolerated in Part A for 28-days, this study will then move to enrolling Part B to evaluate the safety and tolerability of rHSC-DIPGVax and BALSTILIMAB in combination with ZALIFRELIMAB at two dose levels for a total therapy duration of one year or twenty-seven cycles, whichever occurs first.

Advancement from Part A to Part B and dose escalation in Part B will follow a conservative 3+3 design. The dose limiting toxicity (DLT) monitoring period will last 28 days (2 cycles) for Part A subjects and 42 days (1 cycle) for Part B. Subjects will be allowed to continue on in Part A for twenty-seven 14-day cycles or nine 42-day cycles in Part B or 1 year of total therapy, whichever comes first.

After the RP2D of ZALIFRELIMAB is determined, Part C, the expansion arm, will enroll further subjects at this dose level to assess futility versus efficacy. All subjects in trial Part C will be monitored for dose limiting toxicities for the duration of their participation in the study to monitor for excess toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with newly diagnosed typical or non-typical, biopsy-proven DIPG or DMG are eligible for study enrollment. Biopsy is not required for subjects with radiographically typical DIPG meeting imaging criteria. Biopsy is required for DMG's and non-radiographically typical DIPG. Histone mutation must be confirmed by pathology report. Radiographically typical DIPG defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons.

  = Subjects ages > or = to 12 months and < or = 18 years ("Lead In", Part A, and Part B require first three patients be > or = to 12 years of age)
* BSA > or = 0.35m2 at the time of study enrollment
* Performance score: Karnofsky >50% of subjects >16 years of age and Lansky > or = 50 for subjects < or = 16 years of age. Subjects who are unable to walk because of paralysis but are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
* Must start radiation therapy within 42 days from date of diagnostic imaging. C1D1 must be within 42 days to 70 days post radiation (6-10 weeks). Patients CANNOT receive temozolomide during radiation
* Corticosteroids should be weaned as tolerated after radiation therapy with the goal of < or = 0.5mg/kg/day for a minimum of 7 days prior to enrollment.
* Subjects must have measurable disease

Exclusion Criteria:

* Patients cannot receive temozolomide during radiation
* Disseminated disease
* Subjects who have received any cancer therapy except for radiation
* Autoimmune or immune disorders
* Active respiratory disorder or infection
* Active viral infection

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Dose limiting toxicities of rHSC-DIPGVax | DLT period of 28 days for rHSC-DIPGVax monotherapy
  Number of DLT's per CTCAE version 5.0 and iRANO guidelines.
Safety and Tolerability: Dose limiting toxicities of rHSC-DIPGVax plus BALSTILIMAB | DLT period of 28 days for Part A
  Number of DLT's per CTCAE version 5.0 and iRANO guidelines.
Safety and Tolerability: Dose limiting toxicities of rHSC-DIPGVax plus BALSTILIMAB and ZALIFRELIMAB | DLT period of 42 days for Part B
  Number of DLT's per CTCAE version 5.0 and iRANO guidelines.

SECONDARY OUTCOMES:
Total number of DLT's for ZALIFRELIMAB at RP2D in combination with rHSC-DIPGVax and BALSTILIMAB | On-going during 1 year of therapy plus 3 month follow up
  Number of DLT's using CTCAE version 5.0 and iRANO guidelines
To evaluate the efficacy of the combination of rHSC-DIPGVax, BALSTILIMAB, and ZALIFRELIMB in pediatric subjects with DIPG and DMG as measured by overall survival at 12 months and time-to-progression as measured from time of diagnostic imaging | On-going during 1 year of therapy plus 3 month follow up
  12 month overall survival
Overall survival at 1 year | On-going during 1 year of therapy
  Overall survival from time of diagnostic imaging to time of death
Time to progression | On-going during 1 year of therapy plus up to 5 years off treatment
  time to progression (from time of diagnostic imaging to time of disease progression)

OTHER OUTCOMES:
To evaluate biologic correlates for immune response in order to assess neo-antigen specific T cell responses | At the end of each cycle (1 cycle = 28 days) fore the first 3 cycles, on day 1 of cycle 6, and at 3 month post treatment follow up
  PBMC immune subsets measured via flow cytometry from peripheral blood samples
To characterize PK profile (Cmax) of BALSTILIMAB as a mAb monotherapy with rHSC-DIPGVax and in mAb combination with ZALIFRELIMAB and rHSC-DIPGVax to assess potential impact on PK exposure and biologic activity in pediatrics | 1 cycle = 28 days; Predose Cycle 1 day 1, 2 hours post dose 1, cycle 1 day 2, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 predose and 2 hours post dose, cycle 4 day 2, cycle 4 day 8, cycle 5 day 1, cycle 10 day 1, cycle 15 day 1, and end of treatment
  peak plasma concentration (Cmax) of BALSTILIMAB AND ZALIFRELIMAB in the blood
To characterize PK profile (AUC) of BALSTILIMAB as a mAb monotherapy with rHSC-DIPGVax and in mAb combination with ZALIFRELIMAB and rHSC-DIPGVax to assess potential impact on PK exposure and biologic activity in pediatrics | 1 cycle = 28 days; Predose Cycle 1 day 1, 2 hours post dose 1, cycle 1 day 2, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 predose and 2 hours post dose, cycle 4 day 2, cycle 4 day 8, cycle 5 day 1, cycle 10 day 1, cycle 15 day 1, and end of treatment
  Area under the plasma concentration versus time curve (AUC) of BALSTILIMAB AND ZALIFRELIMAB in the blood
To evaluate the immunogenicity of BALSTILIMAB as mAb monotherapy with rHSC-DIPGVax and in mAb combination with ZALIFRELIMAB and rHSC-DIPGVax | 1 cycle = 42 days; Predose on cycle 1 day 1, 2 hours post dose 1, cycle 1 day 2, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1 predose and 2 hours post dose, cycle 4 day 2, cycle 4 day 8, cycle 5 day 1, cycle 10 day 1, cycle 15 day 1, and end of treatment
  Assays to assess anti drug antibody levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Plant-Fox, MD, Principal Investigator — Ann and Robert H. Lurie Children's Hospital
Locations (3):
- United States (3):
  - Children's Health Orange County (CHOC), Orange, California
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No